CLINICAL TRIAL: NCT05971745
Title: Accuracy of Pediatric Emergency Medicine Providers in Diagnosing Hip Effusions Using Point of Care Ultrasound
Status: Completed | Type: Observational
Sponsor: Connecticut Children's Medical Center (Other)
Collaborators: Columbia University (Other); Newark Beth Israel Medical Center (Other); Cohen Children's Medical Center (Other); Gold Coast Hospital and Health Service (Other Government); Yale University (Other)
Responsible Party: Principal Investigator, Ruchika Jones, Principal Investigator, Connecticut Children's Medical Center
Other Study IDs: 19-117
Record Dates: First submitted 2023-07-13; First posted 2023-08-02 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Hip Effusion; Septic Arthritis; Transient Synovitis, Hip
Keywords: Point of Care Ultrasound; Hip Effusion; Pediatric Emergency Medicine
MeSH Terms: conditions — Arthritis, Infectious

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine if pediatric emergency medicine providers can accurately diagnose a hip effusion using point-of-care ultrasound (POCUS) compared to radiology ultrasound (RADUS).

DETAILED DESCRIPTION:
The purpose of this study is to determine that the accuracy of trained pediatric emergency medicine providers to diagnose hip effusion using point-of-care ultrasound (POCUS) is non-inferior to the reference standard of radiology ultrasound (RADUS). Additionally, the investigators seek to compare how POCUS performs against other clinical tests or investigations for the diagnosis of septic arthritis. The investigators hypothesize that trained EM providers will be able to diagnose hip effusions with high (>90%) accuracy compared to studies conducted by the Department of Radiology.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or younger
* Clinical presentation necessitating hip ultrasonography as determined by the evaluating clinician
* Study physician available at the time of presentation to ED
* Patient or legal guardian provides consent

Exclusion Criteria:

* Children who present when a study physician is not available or those for whom consent is not given.
* Children who have had hip ultrasound imaging prior to their ED visit. Children with prior hip/pelvis x-rays will not be excluded.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The target population are children 18 years and younger presenting to the Emergency Department at Connecticut Children's Medical Center with a chief complaint that necessitates hip ultrasonography as determined by the physician caring for the patient at the time of the visit. Those presenting during the study period of October 2019-December 2023 will be recruited. This is a multi-center, international study that will also be conducted in the Pediatric Emergency Departments at the following institutions: Connecticut Children's, Cohen Children's Medical Center, New York-Presbyterian / Columbia University Medical Center, Yale New Haven Hospital, Newark Beth Israel Medical Center, and Gold Coast Hospital (Queensland, Australia).
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
The presence or absence of a hip effusion. | From the time the point-of-care ultrasound is performed by the physician during the emergency department visit through study completion, average of 2 years.
  The presence or absence of an effusion as determined by the pediatric emergency medicine physician performing the point-of-care-ultrasound study on both the affected and unaffected sides (i.e. right hip and left hip).
The presence of absence of a hip effusion. | From the time the radiologist reviews the ultrasound as performed by the radiology technician during the emergency department visit, through study completion, average of 2 years.
  The presence or absence of an effusion as determined by the Radiologist on both the affected and unaffected sides.

SECONDARY OUTCOMES:
The size of the effusion. | From the time the point-of-care ultrasound is performed by the physician during the emergency department visit to study completion, average of 2 years
  As measured by the pediatric emergency medicine provider in millimeters.
The location of the measurement of the effusion. | Upon chart review: between the time the measurement was obtained in the emergency department up to six weeks later when the chart is reviewed by primary investigator.
  Pediatric emergency medicine physicians will measure an effusion at two designated locations. One location is based off of current published literature whereas the second is to provide a comparison to determine if the exact location alters the final diagnosis (effusion or no effusion). Investigators will determine whether the location along the angle of the neck affects the measurement obtained when compared with the current standard practice of measuring fluid along the widest part of the femoral neck.

OTHER OUTCOMES:
Number of point-of-care ultrasound studies performed by PEM providers that have a different final diagnosis when compared to radiology ultrasound. | Upon chart review: between the time the measurement was obtained in the emergency department up to six weeks later when the chart is reviewed by primary investigator.
  Investigators will compare the final diagnosis (hip effusion or no hip effusion) between point-of-care-ultrasound and radiology ultrasound to determine the number of discrepancies between the groups.
Association between point-of-care ultrasound and Kocher score (0-4). | Upon chart review: between the time the measurement was obtained in the emergency department up to six weeks later when the chart is reviewed by primary investigator.
  Investigators will determine if the addition of ultrasonography results coupled with Kocher score (0-4; increased risk of septic arthritis with higher scores), which includes laboratory markers, increases the likelihood of septic arthritis.

CONTACTS AND LOCATIONS:
Overall Officials: Ruchika M Jones, MD, MS, Principal Investigator — Connecticut Children's
Locations (6):
- United States (5):
  - Ruchika M Jones, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Cohen Children's Medical Center, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
- Gold Coast Hospital and Health Service, Southport, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Yes
Each study site will enter data into Redcap hosted by the lead site, Connecticut Children's. Data will be available for review and combined by Connecticut Children's investigators for data analysis. Each participating site has completed a data use agreement with the lead site agreeing to this plan.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Shared as patients are seen throughout the course of the study.
Access Criteria: Only the designated study investigator at each participating site will have Redcap access for purposes of data entry only. Primary investigators at the lead site will have access to the combined data set for data analyses.

REFERENCES:
- [Result] Caird MS, Flynn JM, Leung YL, Millman JE, D'Italia JG, Dormans JP. Factors distinguishing septic arthritis from transient synovitis of the hip in children. A prospective study. J Bone Joint Surg Am. 2006 Jun;88(6):1251-7. doi: 10.2106/JBJS.E.00216. PMID 16757758
- [Result] Kocher MS, Zurakowski D, Kasser JR. Differentiating between septic arthritis and transient synovitis of the hip in children: an evidence-based clinical prediction algorithm. J Bone Joint Surg Am. 1999 Dec;81(12):1662-70. doi: 10.2106/00004623-199912000-00002. PMID 10608376
- [Result] Klein DM, Barbera C, Gray ST, Spero CR, Perrier G, Teicher JL. Sensitivity of objective parameters in the diagnosis of pediatric septic hips. Clin Orthop Relat Res. 1997 May;(338):153-9. doi: 10.1097/00003086-199705000-00022. PMID 9170376
- [Result] Del Beccaro MA, Champoux AN, Bockers T, Mendelman PM. Septic arthritis versus transient synovitis of the hip: the value of screening laboratory tests. Ann Emerg Med. 1992 Dec;21(12):1418-22. doi: 10.1016/s0196-0644(05)80052-6. PMID 1443834
- [Result] Fabry G, Meire E. Septic arthritis of the hip in children: poor results after late and inadequate treatment. J Pediatr Orthop. 1983 Sep;3(4):461-6. doi: 10.1097/01241398-198309000-00008. PMID 6630490
- [Result] Lunseth PA, Heiple KG. Prognosis in septic arthritis of the hip in children. Clin Orthop Relat Res. 1979 Mar-Apr;(139):81-5. PMID 455855
- [Result] Hallel T, Salvati EA. Septic arthritis of the hip in infancy: end result study. Clin Orthop Relat Res. 1978 May;(132):115-28. PMID 307996
- [Result] Bennett OM, Namnyak SS. Acute septic arthritis of the hip joint in infancy and childhood. Clin Orthop Relat Res. 1992 Aug;(281):123-32. PMID 1499198
- [Result] Kocher MS, Mandiga R, Zurakowski D, Barnewolt C, Kasser JR. Validation of a clinical prediction rule for the differentiation between septic arthritis and transient synovitis of the hip in children. J Bone Joint Surg Am. 2004 Aug;86(8):1629-35. doi: 10.2106/00004623-200408000-00005. PMID 15292409
- [Result] Cruz AI Jr, Anari JB, Ramirez JM, Sankar WN, Baldwin KD. Distinguishing Pediatric Lyme Arthritis of the Hip from Transient Synovitis and Acute Bacterial Septic Arthritis: A Systematic Review and Meta-analysis. Cureus. 2018 Jan 25;10(1):e2112. doi: 10.7759/cureus.2112. PMID 29581924
- [Result] Plumb J, Mallin M, Bolte RG. The role of ultrasound in the emergency department evaluation of the acutely painful pediatric hip. Pediatr Emerg Care. 2015 Jan;31(1):54-8; quiz 59-61. doi: 10.1097/PEC.0000000000000332. PMID 25560622
- [Result] Laine JC, Denning JR, Riccio AI, Jo C, Joglar JM, Wimberly RL. The use of ultrasound in the management of septic arthritis of the hip. J Pediatr Orthop B. 2015 Mar;24(2):95-8. doi: 10.1097/BPB.0000000000000134. PMID 25588046
- [Result] Ehrendorfer S, LeQuesne G, Penta M, Smith P, Cundy P. Bilateral synovitis in symptomatic unilateral transient synovitis of the hip: an ultrasonographic study in 56 children. Acta Orthop Scand. 1996 Apr;67(2):149-52. doi: 10.3109/17453679608994660. PMID 8623569
- [Result] Yabunaka K, Ohue M, Morimoto N, Kitano N, Shinohara K, Takamura M, Gotanda T, Sanada S. Sonographic measurement of transient synovitis in children: diagnostic value of joint effusion. Radiol Phys Technol. 2012 Jan;5(1):15-9. doi: 10.1007/s12194-011-0128-z. Epub 2011 Jul 12. PMID 21748477
- [Result] Agarwal A, Aggarwal AN. Bone and Joint Infections in Children: Septic Arthritis. Indian J Pediatr. 2016 Aug;83(8):825-33. doi: 10.1007/s12098-015-1816-1. Epub 2015 Jul 21. PMID 26189923
- [Result] Vieira RL, Levy JA. Bedside ultrasonography to identify hip effusions in pediatric patients. Ann Emerg Med. 2010 Mar;55(3):284-9. doi: 10.1016/j.annemergmed.2009.06.527. Epub 2009 Aug 20. PMID 19695738
- [Result] Luhmann SJ, Jones A, Schootman M, Gordon JE, Schoenecker PL, Luhmann JD. Differentiation between septic arthritis and transient synovitis of the hip in children with clinical prediction algorithms. J Bone Joint Surg Am. 2004 May;86(5):956-62. doi: 10.2106/00004623-200405000-00011. PMID 15118038